CLINICAL TRIAL: NCT07305688
Title: Climate Anxiety in a Young Population at Risk of Suicide
Acronym: Anx-RS
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Esquirol (Other)
Collaborators: Mireille BELLE MBOU (Unknown); Emma BEAU (Unknown)
Responsible Party: Principal Investigator, Bertrand Olliac, Professor, Centre Hospitalier Esquirol
Other Study IDs: 2025-A00139-40
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; Suicidal Ideation; Mental Health Issue; Environmental Exposure
Keywords: Eco-anxiety; Anxiety disorders; Suicide risk; Mental health; Young adults
MeSH Terms: conditions — Anxiety Disorders; Suicidal Ideation; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young Population at Suicide Risk: Adolescents and young adults aged 16-24 years, recruited from emergency, inpatient, and outpatient psychiatry units at Esquirol Hospital Center (France). Participants complete standardized questionnaires assessing climate change anxiety (CCAS-FR), suicidal ideation and behavior (C-SSRS), and general anxiety (STAI-C or STAI-Y).
  Interventions: Other: Columbia Suicide Severity Rating Scale; Other: Climate Change Anxiety Scale - French version; Other: State-Trait Anxiety Inventory, French version; Other: Socio demographic profil

INTERVENTIONS:
Other: Columbia Suicide Severity Rating Scale — Standardized tool for evaluating suicidal ideation and behavior. Measures severity and intensity of suicidal thoughts and actions.
Other: Climate Change Anxiety Scale - French version — 22-item self-report questionnaire assessing cognitive, emotional, functional, and pro-environmental dimensions of climate change-related anxiety.
Other: State-Trait Anxiety Inventory, French version — 40-item self-report inventory measuring both state and trait anxiety levels.
Other: Socio demographic profil — Collects demographic and background variables such as age, gender, education level and living conditions.

SUMMARY:
Background Climate change has become a major source of concern, particularly among younger generations who are facing the progressive degradation of ecosystems, loss of biodiversity, and alarming environmental information disseminated through the media. The direct perception of climate-related disruptions has been shown to engender a profound sense of helplessness and loss. This distress, termed eco-anxiety, is characterised by feelings of fear, sadness and guilt regarding the planet's future.

In a context where there has been a marked increase in suicidal thoughts and attempts among young people over the past decade, it is essential to explore the psychological manifestations of eco-anxiety within this vulnerable population. The paucity of studies investigating this association underscores the significance of the present research.

Principal objective The present study aims to examine the relationship between climate anxiety and suicidal risk among young people aged 16 to 24 years.

Methods This observational, cross-sectional, and multicentre study will be conducted at the Esquirol Hospital Center and the Mother and Child Hospital of Limoges, as well as at the Departmental Hospital Center La Candélie in Agen.

The study will encompass 108 young participants aged between 16 and 24 years, who are either hospitalised or receiving outpatient psychiatric care.

Each participant will be required to complete one clinician-administered assessment, namely the Columbia Suicide Severity Rating Scale (C-SSRS), and two self-report questionnaires: the Climate Change Anxiety Scale - French version (CCAS-FR) and the State-Trait Anxiety Inventory (STAI-Y).

Furthermore, a sociodemographic questionnaire will be administered in order to collect information regarding the subjects' age, sex, education level, living conditions, and psychiatric history.

Perspectives It is hypothesised that there is a positive association between climate anxiety and suicidal risk, with the most eco-anxious participants showing higher C-SSRS scores. It is further predicted that eco-anxiety will correlate with elevated levels of state and trait anxiety, with the potential for modulating this relationship by sociodemographic factors, including gender.

Expected benefits This study will contribute to a better understanding of the psychological impacts of climate change on young people and help identify the most vulnerable profiles. The findings could support suicide prevention strategies, guide the development of specific therapeutic tools for eco-anxious youth, and foster future longitudinal research on the evolution of these conditions and their comorbidities

DETAILED DESCRIPTION:
The Anx-RS France study investigates the association between climate change-related anxiety (eco-anxiety) and suicidal ideation among young people aged 16 to 24 years in France. Growing evidence suggests that climate change may contribute to psychological distress and feelings of hopelessness in younger generations. However, data on the link between eco-anxiety and suicide risk in this age group remain limited.

This is an observational, cross-sectional study including 108 participants recruited from university settings and the general population in France. Eligible participants are aged 16-24 years, fluent in French, and provide informed consent (parental consent is obtained for minors). Participants will be excluded if they have a health condition that prevents them from understanding or completing the study questionnaires. This includes major sensory impairments (e.g., deafness, blindness), severe psychiatric disorders affecting cognition or communication (e.g., acute psychosis, pervasive developmental disorder, confusional state), or current hospitalization in specialized psychiatric units for severe mental illness.

Participants complete a self-administered online survey composed of three validated instruments:

* Climate Change Anxiety Scale (CCAS) - measuring anxiety, rumination, and functional impairment related to climate change.
* State-Trait Anxiety Inventory (STAI-T/Y) - assessing general trait anxiety levels.
* Columbia Suicide Severity Rating Scale (C-SSRS) - evaluating suicidal ideation and behavior.

Descriptive analyses will estimate the prevalence and intensity of climate-related anxiety. Correlational and multivariate analyses will assess the association between eco-anxiety (CCAS) and suicidal ideation (C-SSRS), adjusting for general anxiety levels (STAI-T/Y).

The results will improve understanding of how climate-related distress affects mental health and suicide risk among young people in France, and support prevention strategies and mental-health policy adaptation to emerging environmental stressors.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, boys and girls ;
* Aged between 16 and 24;
* Participants seen in adult or pediatric emergency departments, hospitalised in adult psychiatry or in child and adolescent psychiatry, or seen in outpatient consultation at Esquirol Hospital Center ;
* Affiliated with a social security scheme or entitled to coverage under one ;
* Having received full information about the study and having co-signed, together with the investigator, an informed consent form to participate in the study.
* For minor participants: the consent to participate in the study must be signed by the holder(s) of parental authority, and the minor's assent will also be required.

Exclusion Criteria:

* Participants will not be included in the study if their health condition is incompatible with understanding or completing the questionnaires used. This includes, in particular ;
* Any chronic somatic pathology or major sensory impairment (for example : deafness or blindness) preventing reading, comprehension or communication with healthcare professionals ;
* Any severe psychiatric pathology that significantly impairs cognitive or communication abilities, such as acute psychotic disorders, pervasive developmental disorders or confusional states ;
* Participants hospitalised in units specialising in severe psychiatric disorders with major impairment of cognitive functions.
* Adults under legal protection, in accordance with article L 1121-8 of the Public Health Code ;
* Insufficient command of the French language

Ages: 16 Years to 24 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study population consists of 108 adolescents and young adults aged 16 to 24 years, recruited within the Esquirol Hospital Center (France). Participants are approached in adult and pediatric emergency departments, adult psychiatry, and child and adolescent psychiatry units, as well as during outpatient consultations.
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-01-16 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Climate Change Anxiety Score | 10 min
  Global score from the 13-item French version of the Climate Change Anxiety Scale (CCAS-FR), obtained by summing the cognitive, emotional, and functional disturbance subscales. Higher scores indicate greater levels of climate change-related anxiety.
  Score ranges 13 to 65
Suicide Risk Score | 10 min
  Overall score of suicidal ideation and behavior assessed using the Columbia Suicide Severity Rating Scale (C-SSRS). Higher scores indicate greater suicide risk Score ranges from 2 to 25.

SECONDARY OUTCOMES:
Extended Dimensions of Climate Change Anxiety | 10 min
  Subdimension scores from the extended version of the CCAS-FR, assessing cognitive, emotional, and functional disturbances, as well as direct or indirect experience of climate change and pro-environmental behaviors.
State and Trait Anxiety Scores | 20 min
  Anxiety levels measured using the State-Trait Anxiety Inventory (STAI). The STAI-C is used for participants aged 16-17 years, and the STAI-Y for those aged 18-24 years. Separate state and trait anxiety scores will be analyzed Score ranges 20 to 80

IPD SHARING:
Plan to Share IPD: No